CLINICAL TRIAL: NCT01172951
Title: A Nutrigenomics Study of Post-prandial Metabolic Responses in Individuals of Varying Body Weight: An Assessment of the Body's Response to Meals Containing Different Levels of Fat and Carbohydrate
Brief Title: Nutrigenomics Investigation of the Body's Metabolic Response to 2 Different Meal Challenges
Acronym: MECHE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College Dublin (Other)
Responsible Party: Prof. Mike Gibney, Institute of Food and Health, University College Dublin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: LS-08-43-GR; DAF- HRB (Ireland) (Other Grant/Funding Number: 07FHRIUCD1)
Record Dates: First submitted 2010-07-29; First posted 2010-07-30 (Estimated); Last update posted 2011-01-11 (Estimated); Status verified 2011-01

CONDITIONS: Healthy Subjects
Keywords: Post-prandial; Nutrigenomic; Test meal; Oral glucose tolerance test; Oral lipid tolerance test
MeSH Terms: interventions — Glucose Tolerance Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- OGTT-OGTT-Physical tests (Active Comparator): 2 successive Oral Glucose Tolerance Tests followed by a physical tests session
  Interventions: Other: Oral glucose tolerance test
- OLTT-OLTT-Physical tests (Active Comparator): 2 successive Oral Lipid Tolerance Tests followed by a physical test session
  Interventions: Other: Oral lipid tolerance test
- OGTT-OLTT-Physical tests (Active Comparator): Oral glucose tolerance test followed by an oral lipid tolerance test (or vice-versa) followed by a physical tests session
  Interventions: Other: Oral glucose tolerance test; Other: Oral lipid tolerance test

INTERVENTIONS:
Other: Oral glucose tolerance test — 75g anhydrous glucose powder mixed with 100mls water
  Arms: OGTT-OGTT-Physical tests; OGTT-OLTT-Physical tests
Other: Oral lipid tolerance test — 150ml drink composed of 2 commercially available high fat products
  Arms: OGTT-OLTT-Physical tests; OLTT-OLTT-Physical tests

SUMMARY:
The purpose of this study is to investigate the biological response to a metabolic stress, given in the form of a high carbohydrate or fat meal in normal weight, overweight and obese individuals and to further explore these responses using novel metabolomic, proteomic, transcriptomic and genotyping techniques.

DETAILED DESCRIPTION:
The most recent statistics from the Department of Health in Ireland (2005) indicate that the leading causes of death are those in which nutrition can play a key preventative role. The proposed study will provide information on the metabolic stress from varying body weight overlaid by the additional metabolic stress of a test-meal challenge, in this case being delivered in the form of an oral glucose tolerance test (OGTT) and oral lipid tolerance test (OLTT), standard metabolic challenges in post-prandial research. Previous studies assessing metabolic risk factors associated with a disease have typically focused on information collected from individuals in a fasting state only. However, it is equally important to assess how the body responds when stressed. Employing an acute high fat or carbohydrate intake is sufficient to induce a mild stress in which time an individual's unique post-prandial response can be monitored. This study will combine traditional markers (dietary, anthropometric, lifestyle, clinical and physical activity) with nutrigenomics, a tool that attempts to describe the genome-wide influences of nutrition by examining the impact of diet on genes (genomics), mRNA (transcriptomics), proteins (proteomics) and metabolites (metabolomics).

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 60 years
* Not taking medication (other than contraceptive pill/HRT)
* Irish resident and living in Dublin area

Exclusion Criteria:

* Known chronic/infectious disease
* Pregnancy/lactation
* Desire to conceive or lose weight during study
* Athlete

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2008-12; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Comprehensive analysis of the metabolic response to the acute ingestion of fat and glucose loads | 2-5 hours post test meal ingestion

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Gibney, PhD, Principal Investigator — University College Dublin; Donal O'Shea, MD, Principal Investigator — St Vincent's University Hospital, Ireland; Helen Roche, PhD, Principal Investigator — University College Dublin; Lorraine Brennan, PhD, Principal Investigator — University College Dublin; Eileen Gibney, PhD, Principal Investigator — University College Dublin
Locations (2):
- Ireland (2):
  - Institute for Sport and Health, University College Dublin, Dublin
  - St Vincent's University Hospital, Dublin

REFERENCES:
- [Derived] Jackson KG, Li Y, Ryan MF, Gibney ER, Brennan L, Roche HM, Williams CM, Lovegrove JA, Vimaleswaran KS. Association of the tumor necrosis factor-alpha promoter polymorphism with change in triacylglycerol response to sequential meals. Nutr J. 2016 Jul 25;15(1):70. doi: 10.1186/s12937-016-0190-9. PMID 27456841
- [Derived] Matone A, O'Grada CM, Dillon ET, Morris C, Ryan MF, Walsh M, Gibney ER, Brennan L, Gibney MJ, Morine MJ, Roche HM. Body mass index mediates inflammatory response to acute dietary challenges. Mol Nutr Food Res. 2015 Nov;59(11):2279-92. doi: 10.1002/mnfr.201500184. Epub 2015 Sep 22. PMID 26314729
- [Derived] Morris C, O'Grada CM, Ryan MF, Gibney MJ, Roche HM, Gibney ER, Brennan L. Modulation of the lipidomic profile due to a lipid challenge and fitness level: a postprandial study. Lipids Health Dis. 2015 Jul 1;14:65. doi: 10.1186/s12944-015-0062-x. PMID 26123789
- [Derived] Ferguson JF, Ryan MF, Gibney ER, Brennan L, Roche HM, Reilly MP. Dietary isoflavone intake is associated with evoked responses to inflammatory cardiometabolic stimuli and improved glucose homeostasis in healthy volunteers. Nutr Metab Cardiovasc Dis. 2014 Sep;24(9):996-1003. doi: 10.1016/j.numecd.2014.03.010. Epub 2014 Apr 18. PMID 24875672
- [Derived] Wallace M, Morris C, O'Grada CM, Ryan M, Dillon ET, Coleman E, Gibney ER, Gibney MJ, Roche HM, Brennan L. Relationship between the lipidome, inflammatory markers and insulin resistance. Mol Biosyst. 2014 Jun;10(6):1586-95. doi: 10.1039/c3mb70529c. Epub 2014 Apr 9. PMID 24714806
- [Derived] Morris C, Grada CO, Ryan M, Roche HM, De Vito G, Gibney MJ, Gibney ER, Brennan L. The relationship between aerobic fitness level and metabolic profiles in healthy adults. Mol Nutr Food Res. 2013 Jul;57(7):1246-54. doi: 10.1002/mnfr.201200629. Epub 2013 Mar 15. PMID 23505034
- [Derived] Ryan MF, O'Grada CM, Morris C, Segurado R, Walsh MC, Gibney ER, Brennan L, Roche HM, Gibney MJ. Within-person variation in the postprandial lipemic response of healthy adults. Am J Clin Nutr. 2013 Feb;97(2):261-7. doi: 10.3945/ajcn.112.047936. Epub 2013 Jan 2. PMID 23283501
- [Derived] Morris C, O'Grada C, Ryan M, Roche HM, Gibney MJ, Gibney ER, Brennan L. The relationship between BMI and metabolomic profiles: a focus on amino acids. Proc Nutr Soc. 2012 Nov;71(4):634-8. doi: 10.1017/S0029665112000699. Epub 2012 Aug 6. PMID 22863201